CLINICAL TRIAL: NCT00672932
Title: Pilot Study of Raltegravir Augmentation on Persistent Central Nervous System (CNS) Immunoactivation in Treated HIV-1 Patients
Brief Title: Raltegravir Augmentation on Persistent Central Nervous System (CNS) Immunoactivation in Treated HIV-1 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CCRC5004; R01MH062701 (NIH)
Record Dates: First submitted 2008-04-29; First posted 2008-05-06 (Estimated); Results first posted 2013-07-05 (Estimated); Last update posted 2013-07-05 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections
Keywords: raltegravir; central nervous system (CNS); HIV-1; AIDS; cerebrospinal fluid (CSF); immunoactivation; antiretroviral therapy; suppression
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- raltegravir group (Experimental): The raltegravir dosing will be 400mg twice daily by mouth. Subjects will continue all of their regular medications throughout the protocol.
  Interventions: Drug: raltegravir
- No augmented treatment (No Intervention): Subjects randomized not to receive augmented treatment will continue in the study with their regular antiretroviral regimen.

INTERVENTIONS:
Drug: raltegravir — 400 mg two times daily for three months
  Other Names: Isentress
  Arms: raltegravir group

SUMMARY:
This pilot study focuses on the persistence of central nervous system (CNS) immune activation that has been observed in the presence of 'effective' combination antiretroviral therapy (cART). Attention to this issue is based on the fear that chronic CNS immunoactivation can cause indolent brain injury that will eventually compromise brain function as patients survive for years on treatment. A leading hypothesis explaining this continued immunoactivation is that viral replication continues within the brain at a level too low for detection in cerebrospinal fluid (CSF), yet sufficient to stimulate local immunoactivation. Based on this hypothesis, we propose to use augmented treatment with raltegravir to test whether additional suppression of this hypothesized CNS HIV-1 replication will reduce continued CNS immunoactivation.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent.
* Documented HIV-1 infection.
* History of continuous cART treatment (with at least three drugs) for at least 2 years.
* Documentation of 'undetectable' plasma HIV-1 RNA for at least 1 year.
* HIV-1 RNA <50 copies/mL in plasma and CSF at screening visit.

Exclusion Criteria:

* Contraindication to LP (suspicion of CNS mass lesion, bleeding diathesis, etc.).
* Prior experience with raltegravir or contraindication to raltegravir treatment, including medication interactions that might compromise ongoing antiretroviral therapy or treatment of other conditions.
* Active opportunistic infections or neurological diseases.
* Other conditions or treatments likely to interfere with treatment or evaluation.
* Hemoglobin < 10 Gm/dL.
* Pregnant or anticipating pregnancy during study.
* Active substance abuse.
* Subjects taking rifampin, phenytoin, Phenobarbital or other drugs that accelerate raltegravir metabolism and might decrease its tissue concentrations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Price, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Ucsf Ccrc, Sfgh, San Francisco, California, United States

REFERENCES:
- [Result] Dahl V, Lee E, Peterson J, Spudich SS, Leppla I, Sinclair E, Fuchs D, Palmer S, Price RW. Raltegravir treatment intensification does not alter cerebrospinal fluid HIV-1 infection or immunoactivation in subjects on suppressive therapy. J Infect Dis. 2011 Dec 15;204(12):1936-45. doi: 10.1093/infdis/jir667. Epub 2011 Oct 21. PMID 22021620

RESULTS

PARTICIPANT FLOW:
Groups:
- No Augmented Treatment Then Optional Rollover: Subjects randomized not to receive augmented treatment will continue in the study with their regular antiretroviral regimen. After 12 weeks, subjects in this group have the option to rollover into the raltegravir group for 12 weeks.
Period: Overall Study
Arm/Group | Raltegravir Group | No Augmented Treatment Then Optional Rollover
Started | 9 | 9
Completed Initial 12-week Assignment | 9 | 9
Provided Analyzable Blood and CSF Sample | 8 (one subject was censored when pharmacological study showed no drug in plasma or CSF) | 9
Rolled Over to Raltegravir | 0 | 6 (6 subjects randomized to no drug later rolled over to receive raltegravir)
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir Group | No Augmented Treatment | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 52.7 (6.4) | 54.3 (5.3) | 53.9 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in CD8+ T Cell Co-expression of CD38 and HLA-DR
Description: Blood CD8+ T cell activation as indicated by percentage of cells in fresh specimens coexpressing surface CD38 and human leukocyte antigen (HLA)-DR.
Time Frame: three months (Rollover subjects were assessed for a second baseline after the initial 12 week period)
Population: One subject in the raltegravir group was censored when a pharmacological study showed no drug in either plasma (n=9) or CSF. Six subjects randomized to no drug later rolled over to receive raltegravir. Primary analysis treated the rollover subjects as independent and compared 14 intensified to 9 nonintensified subject experiences.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Raltegravir Group | No Augmented Treatment
Number analyzed (Participants) | 14 | 9
percentage of cells | 0.51 (1.03) | 0.66 (1.20)

2. Primary Outcome: Change in CSF Concentrations of Neopterin After 12 Weeks
Description: CSF markers of immuno¬activation and inflammation after 12 weeks compared to baseline.
Time Frame: three months (Rollover subjects were assessed for a second baseline after the initial 12 week period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Raltegravir Group | No Augmented Treatment
Number analyzed (Participants) | 14 | 9
nmol/L | 0.1 (0.3) | 0.3 (1.1)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: 6 subjects who rolled over to treatment after 12 weeks of no treatment were followed for an additional 12 weeks. 1 subject in the Raltegravir group was not included in other analyses because a pharmacological study showed no drug in either plasma or CSF.
Arm/Group | Raltegravir Group | No Augmented Treatment
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/9
Other Adverse Events (participants affected / at risk) | 0/15 | 0/9

LIMITATIONS AND CAVEATS:
The underlying hypothesis might not have actually been addressed because of the particular makeup of the subject group with minimal CNS infection and immunoactivation that left little room to discern a therapeutic effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No